CLINICAL TRIAL: NCT02424643
Title: Improving Survey Procedures for Young Men Who Have Sex With Men in Web-based HIV Prevention: Retention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB00065333a
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Incentive (No Intervention): Participants in this arm will receive no compensation for taking the online survey.
- Monetary Incentive (Experimental): Participants in this arm will receive a $20 Amazon.com incentive for participating in the online survey.
  Interventions: Behavioral: Monetary Incentive
- Altruistic Incentive (Experimental): Participants in this arm will receive altruistic messages throughout the length of the survey in hopes of improving survey completion.
  Interventions: Behavioral: Altruistic Incentive
- Dashboard Incentive (Experimental): Participants in this arm will receive a dashboard at the end of the survey that will compare their data entered into the survey to other participants who have taken the survey. A preview of this dashboard will be shown at the beginning of the survey as a teaser in the hopes to improve survey completion.
  Interventions: Behavioral: Dashboard Incentive

INTERVENTIONS:
Behavioral: Monetary Incentive — $20 Amazon.com gift card
  Arms: Monetary Incentive
Behavioral: Altruistic Incentive — A preliminary statement of the importance of participation, and periodic "inspirational" messages throughout the length of the survey emphasizing the value to men's health by completing the survey
  Arms: Altruistic Incentive
Behavioral: Dashboard Incentive — A sample "dashboard" will compare data subjects enter in their survey to the data already collected from other men who have taken the survey. For the dashboard, men who complete the survey will be shown how their own reported data about certain topics compared to other men's data.
  Arms: Dashboard Incentive

SUMMARY:
The purpose of this study is to test the efficacy of alternative methods to improve survey completion.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are the risk population most heavily impacted by HIV in the United States by any measure; in 2009, at least 61% of new HIV infections were estimated to have occurred in MSM. MSM are experiencing an increase in HIV transmission that has been occurring since at least 1990, and accelerated in multiple North American and European countries from 2000-2005. The expansion of the HIV epidemic has been proposed to be attributable, in part, to the extent to which the internet has facilitated sexual connectivity among MSM.

Researchers have attempted to reach MSM for HIV prevention research and intervention on the internet. In the past 10 years, there has been a proliferation of internet surveys and HIV research studies among men who have sex with men that utilize the internet for data collection and, in some cases, the delivery of HIV prevention content. The development of internet-based interventions has been recently identified as especially promising because of its potential for scalability. However, there are also important limitations to internet-based data collections and prevention studies. The most important of these relate to representativeness and opportunities to introduce bias to data collections and differences in access to and use of internet among different subgroups of MSM. Equally important, although less discussed, are the unique ethical and human research protections challenges posed by online sexual health prevention studies.

The investigators will conduct an experiment to improve knowledge of how to conduct internet-based HIV prevention research with MSM in ways that decrease biases in data collections. The design will consist of a randomized controlled trials of MSM recruited online. A total of 1000 MSM will be enrolled to determine how to best improve retention in online surveys.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18 to 34 years
* have had sex with another man in the past 12 months

Exclusion Criteria:

* female or transgender
* younger than 18 years of age
* older than 34 years of age
* have not had sex with another man in the past 12 months.

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1131 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of survey completed before dropping out. | At baseline survey
  We expect that the average participant will complete 40 screens of survey in about 45 minutes. Based on historical data, about 75% of participants will complete all screens. Analyses will take a time-to-event approach and hazard of discontinuing survey will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Rollins School of Public Health, Emory University, Atlanta, Georgia, United States